CLINICAL TRIAL: NCT00278889
Title: A Study to Compare the Efficacy of AZD2171 in Combination With 5-fluorouracil, Leucovorin, and Oxaliplatin (FOLFOX) and the Efficacy of Bevacizumab in Combination With FOLFOX in the Second-line Treatment of Patients With Metastatic Colorectal Cancer
Brief Title: Second Line ColoRectal Cancer Therapy in Combination With Combination of FOL- Folinic Acid(Leucovorin), F - Fluorouracil and OX - Oxaliplatin (FOLFOX)
Acronym: HORIZON I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8480C00041; EUDRACT number 2005-003443-31; HORIZON I
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Results first posted 2012-10-24 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; phase II; metastatic colorectal cancer; AZD2171; RECENTIN
MeSH Terms: conditions — Colorectal Neoplasms | interventions — cediranib; Fluorouracil; Leucovorin; Oxaliplatin; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Bevacizumab + FOLFOX
  Interventions: Drug: 5-fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Bevacizumab
- 2 (Experimental): AZD2171 + FOLFOX
  Interventions: Drug: AZD2171; Drug: 5-fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: AZD2171 — oral tablet
  Other Names: cediranib; RECENTIN™
  Arms: 2
Drug: 5-fluorouracil — intravenous infusion
  Other Names: 5-FU
Drug: Leucovorin — intravenous infusion
Drug: Oxaliplatin — intravenous infusion
  Other Names: Eloxatin®
Drug: Bevacizumab — intravenous infusion
  Other Names: Avastin®
  Arms: 1

SUMMARY:
The primary purpose of this study is to compare the efficacy of AZD2171 in combination with FOLFOX to the efficacy of bevacizumab in combination with FOLFOX, in the second-line treatment of patients with metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of colon or rectal cancer,
* Received prior systemic therapy for cancer,
* Cancer must have progressed during or after first treatment

Exclusion Criteria:

* Prior treatment with a VEGF inhibitor,
* Poorly controlled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, Study Director — AstraZeneca
Locations (43):
- Austria (3):
  - Research Site, Innsbruck
  - Research Site, Vienna
  - Research Site, Wels
- Belgium (5):
  - Research Site, Bonheiden
  - Ressearch Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
- Canada (7):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Czechia (4):
  - Research Site, Chomutov
  - Research Site, Nová Ves pod Pleší
  - Research Site, Pardubice
  - Research Site, Prague
- France (2):
  - Research Site, Montpellier
  - Research Site, Saint-Herblain
- Germany (7):
  - Research Site, Berlin
  - Research Site, Freiburg im Breisgau
  - Research Site, Halle
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, München
  - Research Site, Stuttgart
- Italy (5):
  - Research Site, Genova
  - Research Site, La Torretta
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Rozzano
- Spain (5):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Valencia
  - Research Site, Zaragoza
- United Kingdom (5):
  - Research Site, Glasgow
  - Research Site, Ipswich
  - Research Site, Maidstone
  - Research Site, Newcastle upon Tyne
  - Research Site, Sutton

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFOX + Cediranib 20 mg: FOLFOX + Cediranib 20 mg
- FOLFOX + Cediranib 30 mg: FOLFOX + Cediranib 30 mg
- FOLFOX + Bevacizumab 10 mg/kg: FOLFOX + Bevacizumab 10 mg/kg
Period: Overall Study
Arm/Group | FOLFOX + Cediranib 20 mg | FOLFOX + Cediranib 30 mg | FOLFOX + Bevacizumab 10 mg/kg
Started | 73 (Randomised) | 74 (Randomised) | 68 (Randomised)
Overall Survival Analysis | 16 (Ongoing at data cut-off for OS analysis (30 January 2009)) | 20 (Ongoing at data cut-off for OS analysis (30 January 2009)) | 19 (Ongoing at data cut-off for OS analysis (30 January 2009))
Completed | 48 (Ongoing at data cut-off for PFS analysis (November 2007)) | 47 (Ongoing at data cut-off for PFS analysis (November 2007)) | 48 (Ongoing at data cut-off for PFS analysis (November 2007))
Not Completed | 25 | 27 | 20
Not completed — Withdrawal by Subject | 0 | 5 | 3
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Death | 24 | 21 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOLFOX + Cediranib 20 mg | FOLFOX + Cediranib 30 mg | FOLFOX + Bevacizumab 10 mg/kg | Total
Number analyzed (Participants) | 71 | 73 | 66 | 210
Age Continuous [Mean (Standard Deviation); unit: Years]
  Age | 63.9 (8.7) | 63.5 (9.6) | 61.8 (10.6) | 63.07 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 27 | 75
  Male | 49 | 47 | 39 | 135

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Number of months from randomisation to the earlier date of objective progression or death
Time Frame: Randomisation to data cut-off date of November 2007
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | FOLFOX + Cediranib 20 mg | FOLFOX + Cediranib 30 mg | FOLFOX + Bevacizumab 10 mg/kg
Number analyzed (Participants) | 71 | 73 | 66
Months | 5.8 [3.9 to 8.9] | 7.2 [4.6 to 8.8] | 7.8 [5.3 to 10.8]

2. Secondary Outcome: Objective Response Rate
Description: Per RECIST Criteria (V1.0) and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >= ##% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  Confirmed Partial Response (PR) or Complete Response (CR) as defined by RECIST.
Time Frame: Randomisation to data cut-off date of November 2007
Measure: Number; unit: Participants
Arm/Group | FOLFOX + Cediranib 20 mg | FOLFOX + Cediranib 30 mg | FOLFOX + Bevacizumab 10 mg/kg
Number analyzed (Participants) | 71 | 73 | 66
Participants | 13 | 14 | 18

3. Secondary Outcome: Overall Survival
Description: Number of months from randomisation to the date of death from any cause
Time Frame: Randomisation to data cut-off date of 30 January 2009
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | FOLFOX + Cediranib 20 mg | FOLFOX + Cediranib 30 mg | FOLFOX + Bevacizumab 10 mg/kg
Number analyzed (Participants) | 71 | 73 | 66
Months | 14.3 [8.6 to 26.4] | 16.8 [9.4 to 31.1] | 19.6 [12.1 to 27.1]

4. Secondary Outcome: Quality Of Live(QOL) : Time to Worsening of Tissue Oxygen Index (TOI)
Description: Time when a sustained clinically important deterioration in TOI has been recorded: derived from the FACT-C questionnaires
Time Frame: Randomisation to data cut-off date of November 2007
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | FOLFOX + Cediranib 20 mg | FOLFOX + Cediranib 30 mg | FOLFOX + Bevacizumab 10 mg/kg
Number analyzed (Participants) | 64 | 67 | 60
Days | 63 [39 to 143] | 74 [35 to 218] | 87 [56 to 225]

5. Secondary Outcome: QOL: Time to Worsening of Treatment-free Survival (TFS)
Description: Time when a sustained clinically important deterioration in TFS has been recorded: derived from the Functional Assessment of Cancer Therapy-Colorectal (FACT-C) questionnaires
Time Frame: Randomisation to data cut-off date of November 2007
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | FOLFOX + Cediranib 20 mg | FOLFOX + Cediranib 30 mg | FOLFOX + Bevacizumab 10 mg/kg
Number analyzed (Participants) | 63 | 67 | 59
Days | 98 [43 to 171] | 112 [54 to 218] | 147 [61 to 231]

6. Secondary Outcome: QOL: Time to Worsening of Clear Cell Sarcoma (CCS)
Description: Time when a sustained clinically important deterioration in CCS has been recorded: derived from the FACT-C questionnaires
Time Frame: Randomisation to data cut-off date of November 2007
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | FOLFOX + Cediranib 20 mg | FOLFOX + Cediranib 30 mg | FOLFOX + Bevacizumab 10 mg/kg
Number analyzed (Participants) | 64 | 67 | 60
Days | 84 [41 to 159] | 74 [35 to 224] | 87 [56 to 188]

7. Secondary Outcome: QOL: Time to Worsening of FACT Colorectal Cancer Symptom Index(FCSI)
Description: as for outcome 6
Time Frame: Randomisation to data cut-off date of November 2007
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | FOLFOX + Cediranib 20 mg | FOLFOX + Cediranib 30 mg | FOLFOX + Bevacizumab 10 mg/kg
Number analyzed (Participants) | 70 | 69 | 60
Days | 106 [51 to 163] | 92 [35 to 221] | 155 [56 to 232]

ADVERSE EVENTS:
Arm/Group | FOLFOX + Cediranib 20 mg | FOLFOX + Cediranib 30 mg | FOLFOX + Bevacizumab 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 30/73 | 39/74 | 29/68
Other Adverse Events (participants affected / at risk) | 69/73 | 73/74 | 66/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | FOLFOX + Cediranib 20 mg (N=73) | FOLFOX + Cediranib 30 mg (N=74) | FOLFOX + Bevacizumab 10 mg/kg (N=68)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0/70 | 1/73 | 0/66
Granulocytopenia (Blood and lymphatic system disorders) | 1/70 | 0/73 | 0/66
Neutropenia (Blood and lymphatic system disorders) | 0/70 | 0/73 | 1/66
Thrombocytopenia (Blood and lymphatic system disorders) | 1/70 | 1/73 | 0/66
Atrial Fibrillation (Cardiac disorders) | 1/70 | 0/73 | 0/66
Blindness (Eye disorders) | 0/70 | 1/73 | 0/66
Abdominal Pain (Gastrointestinal disorders) | 4/70 | 0/73 | 3/66
Diarrhoea (Gastrointestinal disorders) | 2/70 | 3/73 | 3/66
Small Intestinal Obstruction (Gastrointestinal disorders) | 3/70 | 0/73 | 1/66
Intestinal Obstruction (Gastrointestinal disorders) | 0/70 | 1/73 | 2/66
Stomatitis (Gastrointestinal disorders) | 0/70 | 2/73 | 0/66
Abdominal Symptom (Gastrointestinal disorders) | 0/70 | 0/73 | 1/66
Colitis (Gastrointestinal disorders) | 0/70 | 0/73 | 1/66
Colonic Obstruction (Gastrointestinal disorders) | 1/70 | 0/73 | 0/66
Constipation (Gastrointestinal disorders) | 0/70 | 1/73 | 0/66
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0/70 | 1/73 | 0/66
Gastrointestinal Obstruction (Gastrointestinal disorders) | 0/70 | 0/73 | 1/66
Gastrointestinal Toxicity (Gastrointestinal disorders) | 0/70 | 1/73 | 0/66
Ileus (Gastrointestinal disorders) | 1/70 | 1/73 | 1/66
Ileus Paralytic (Gastrointestinal disorders) | 0/70 | 1/73 | 0/66
Large Intestine Perforation (Gastrointestinal disorders) | 0/70 | 0/73 | 1/66
Proctalgia (Gastrointestinal disorders) | 0/70 | 0/73 | 1/66
Small Intestinal Perforation (Gastrointestinal disorders) | 1/70 | 0/73 | 0/66
Subileus (Gastrointestinal disorders) | 1/70 | 1/73 | 1/66
Vomiting (Gastrointestinal disorders) | 0/70 | 1/73 | 0/66
Asthenia (General disorders) | 0/70 | 3/73 | 0/66
Pyrexia (General disorders) | 1/70 | 2/73 | 2/66
Fatigue (General disorders) | 0/70 | 1/73 | 0/66
Infusion Site Extravasation (General disorders) | 1/70 | 0/73 | 0/66
Malaise (General disorders) | 1/70 | 0/73 | 0/66
Non-Cardiac Chest Pain (General disorders) | 0/70 | 0/73 | 1/66
Sudden Cardiac Death (General disorders) | 0/70 | 1/73 | 0/66
Bile Duct Stone (Hepatobiliary disorders) | 1/70 | 0/73 | 0/66
Hepatic Failure (Hepatobiliary disorders) | 0/70 | 0/73 | 1/66
Drug Hypersensitivity (Immune system disorders) | 0/70 | 1/73 | 1/66
Infection (Infections and infestations) | 0/70 | 0/73 | 2/66
Urinary Tract Infection (Infections and infestations) | 0/70 | 0/73 | 2/66
Bronchitis (Infections and infestations) | 0/70 | 0/73 | 1/66
Catheter Related Infection (Infections and infestations) | 0/70 | 0/73 | 1/66
Central Line Infection (Infections and infestations) | 0/70 | 1/73 | 1/66
Gastroenteritis (Infections and infestations) | 1/70 | 0/73 | 0/66
Klebsiella Bacteraemia (Infections and infestations) | 0/70 | 0/73 | 1/66
Lobar Pneumonia (Infections and infestations) | 1/70 | 0/73 | 0/66
Lung Infection (Infections and infestations) | 1/70 | 0/73 | 1/66
Pneumonia (Infections and infestations) | 0/70 | 1/73 | 1/66
Respiratory Tract Infection (Infections and infestations) | 1/70 | 0/73 | 0/66
Sepsis (Infections and infestations) | 0/70 | 0/73 | 1/66
Sepsis Syndrome (Infections and infestations) | 1/70 | 0/73 | 0/66
Anastomotic Complication (Injury, poisoning and procedural complications) | 1/70 | 0/73 | 0/66
Anastomotic Ulcer (Injury, poisoning and procedural complications) | 1/70 | 0/73 | 0/66
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0/70 | 1/73 | 0/66
Blood Creatinine Increased (Injury, poisoning and procedural complications) | 1/70 | 0/73 | 0/66
Weight Decreased (Injury, poisoning and procedural complications) | 0/70 | 1/73 | 0/66
Anorexia (Metabolism and nutrition disorders) | 0/70 | 3/73 | 1/66
Dehydration (Metabolism and nutrition disorders) | 1/70 | 2/73 | 1/66
Cachexia (Metabolism and nutrition disorders) | 0/70 | 0/73 | 1/66
Hypokalaemia (Metabolism and nutrition disorders) | 0/70 | 1/73 | 0/66
Back Pain (Musculoskeletal and connective tissue disorders) | 0/70 | 0/73 | 1/66
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0/70 | 1/73 | 0/66
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1/70 | 0/73 | 0/66
Cerebral Infarction (Nervous system disorders) | 0/70 | 1/73 | 0/66
Cerebral Ischaemia (Nervous system disorders) | 0/70 | 1/73 | 0/66
Convulsion (Nervous system disorders) | 0/70 | 1/73 | 0/66
Headache (Nervous system disorders) | 1/70 | 0/73 | 0/66
Somnolence (Nervous system disorders) | 0/70 | 1/73 | 0/66
Confusional State (Psychiatric disorders) | 1/70 | 2/73 | 0/66
Agitation (Psychiatric disorders) | 0/70 | 1/73 | 0/66
Hydronephrosis (Renal and urinary disorders) | 1/70 | 0/73 | 0/66
Renal Failure (Renal and urinary disorders) | 0/70 | 1/73 | 0/66
Ureteric Obstruction (Renal and urinary disorders) | 0/70 | 0/73 | 1/66
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | FOLFOX + Cediranib 20 mg (N=73) | FOLFOX + Cediranib 30 mg (N=74) | FOLFOX + Bevacizumab 10 mg/kg (N=68)
Neutropenia (Blood and lymphatic system disorders) | 37/70 | 32/73 | 29/66
Thrombocytopenia (Blood and lymphatic system disorders) | 26/70 | 29/73 | 15/66
Leukopenia (Blood and lymphatic system disorders) | 9/70 | 8/73 | 5/66
Anaemia (Blood and lymphatic system disorders) | 7/70 | 7/73 | 5/66
Hypothyroidism (Endocrine disorders) | 2/70 | 5/73 | 1/66
Diarrhoea (Gastrointestinal disorders) | 52/70 | 54/73 | 42/66
Nausea (Gastrointestinal disorders) | 35/70 | 41/73 | 38/66
Stomatitis (Gastrointestinal disorders) | 22/70 | 33/73 | 25/66
Vomiting (Gastrointestinal disorders) | 22/70 | 28/73 | 25/66
Abdominal Pain (Gastrointestinal disorders) | 18/70 | 21/73 | 14/66
Constipation (Gastrointestinal disorders) | 17/70 | 13/73 | 18/66
Abdominal Pain Upper (Gastrointestinal disorders) | 8/70 | 6/73 | 5/66
Dyspepsia (Gastrointestinal disorders) | 7/70 | 4/73 | 5/66
Aphthous Stomatitis (Gastrointestinal disorders) | 1/70 | 1/73 | 6/66
Dysphagia (Gastrointestinal disorders) | 6/70 | 3/73 | 3/66
Flatulence (Gastrointestinal disorders) | 0/70 | 1/73 | 6/66
Rectal Haemorrhage (Gastrointestinal disorders) | 6/70 | 1/73 | 0/66
Dry Mouth (Gastrointestinal disorders) | 3/70 | 5/73 | 1/66
Toothache (Gastrointestinal disorders) | 5/70 | 3/73 | 3/66
Paraesthesia Oral (Gastrointestinal disorders) | 2/70 | 4/73 | 3/66
Proctalgia (Gastrointestinal disorders) | 4/70 | 0/73 | 1/66
Fatigue (General disorders) | 35/70 | 41/73 | 39/66
Asthenia (General disorders) | 17/70 | 16/73 | 9/66
Pyrexia (General disorders) | 13/70 | 13/73 | 15/66
Oedema Peripheral (General disorders) | 2/70 | 3/73 | 5/66
Chills (General disorders) | 4/70 | 3/73 | 3/66
Mucosal Inflammation (General disorders) | 2/70 | 1/73 | 4/66
Drug Hypersensitivity (Immune system disorders) | 4/70 | 2/73 | 5/66
Nasopharyngitis (Infections and infestations) | 4/70 | 5/73 | 7/66
Urinary Tract Infection (Infections and infestations) | 7/70 | 7/73 | 5/66
Bronchitis (Infections and infestations) | 3/70 | 4/73 | 5/66
Weight Decreased (Infections and infestations) | 17/70 | 7/73 | 8/66
Aspartate Aminotransferase Increased (Infections and infestations) | 5/70 | 4/73 | 1/66
Alanine Aminotransferase Increased (Infections and infestations) | 4/70 | 4/73 | 0/66
Anorexia (Metabolism and nutrition disorders) | 29/70 | 24/73 | 29/66
Hypokalaemia (Metabolism and nutrition disorders) | 12/70 | 5/73 | 5/66
Dehydration (Metabolism and nutrition disorders) | 3/70 | 7/73 | 4/66
Decreased Appetite (Metabolism and nutrition disorders) | 4/70 | 5/73 | 4/66
Hypomagnesaemia (Metabolism and nutrition disorders) | 3/70 | 1/73 | 5/66
Back Pain (Musculoskeletal and connective tissue disorders) | 5/70 | 6/73 | 13/66
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4/70 | 10/73 | 8/66
Arthralgia (Musculoskeletal and connective tissue disorders) | 7/70 | 6/73 | 4/66
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5/70 | 3/73 | 6/66
Paraesthesia (Nervous system disorders) | 20/70 | 31/73 | 24/66
Peripheral Sensory Neuropathy (Nervous system disorders) | 20/70 | 17/73 | 25/66
Headache (Nervous system disorders) | 10/70 | 16/73 | 16/66
Neuropathy Peripheral (Nervous system disorders) | 9/70 | 6/73 | 12/66
Dysgeusia (Nervous system disorders) | 11/70 | 9/73 | 10/66
Dysaesthesia (Nervous system disorders) | 4/70 | 2/73 | 7/66
Dizziness (Nervous system disorders) | 6/70 | 4/73 | 4/66
Polyneuropathy (Nervous system disorders) | 6/70 | 3/73 | 4/66
Lethargy (Nervous system disorders) | 5/70 | 0/73 | 1/66
Insomnia (Psychiatric disorders) | 5/70 | 7/73 | 5/66
Anxiety (Psychiatric disorders) | 2/70 | 4/73 | 4/66
Proteinuria (Renal and urinary disorders) | 13/70 | 13/73 | 15/66
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 22/70 | 21/73 | 13/66
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12/70 | 15/73 | 13/66
Cough (Respiratory, thoracic and mediastinal disorders) | 6/70 | 4/73 | 11/66
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8/70 | 10/73 | 6/66
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0/70 | 1/73 | 4/66
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1/70 | 4/73 | 3/66
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 12/70 | 8/73 | 7/66
Alopecia (Skin and subcutaneous tissue disorders) | 6/70 | 8/73 | 10/66
Pruritus (Skin and subcutaneous tissue disorders) | 2/70 | 1/73 | 8/66
Rash (Skin and subcutaneous tissue disorders) | 0/70 | 8/73 | 8/66
Dry Skin (Skin and subcutaneous tissue disorders) | 4/70 | 7/73 | 1/66
Erythema (Skin and subcutaneous tissue disorders) | 0/70 | 4/73 | 2/66
Night Sweats (Skin and subcutaneous tissue disorders) | 4/70 | 0/73 | 1/66
Hypertension (Vascular disorders) | 35/70 | 43/73 | 32/66
Pallor (Vascular disorders) | 0/70 | 4/73 | 1/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a Study Site, or an investigator, requests permission to publish data from this study, any such publication (including oral presentations) is to be agreed with AstraZeneca prior to publication.